CLINICAL TRIAL: NCT01743430
Title: 1. Telerehabilitation on Balance in Subacute Stroke; 2.Telerehabilitation on Balance and Daily Activities in Chronic Stroke; 3. Telerehabilitation on Quality of Life in Chronic Stroke; 4. Telerehabilitation on Satisfaction in Stroke
Brief Title: Development of Smart Holistic Telerehabilitation System: An Application of Stroke Patients- 3 Years Study
Acronym: telerehab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 200809040R
Record Dates: First submitted 2011-10-20; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-11

CONDITIONS: Stroke
Keywords: telerehabilitation; stroke; Berg balance scale; stroke impact scale; mobility
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telerehabilitation (Experimental): telerehabilitation via internet
  Interventions: Other: telerehabilitation
- conventional (No Intervention): conventional therapy

INTERVENTIONS:
Other: telerehabilitation — telerehabilitation for 4 weeks, 2 sessions per week and 30 to 50 minutes per session
  Other Names: physical therapy
  Arms: telerehabilitation

SUMMARY:
Study 1: Background and Purpose-This study were to set up the telerehabilitation program for standing balance training, and to examine the training effects on balance and daily activities in subjects with subacute stroke.The null hypothesis included telerehabilitation balance training were not significantly different from conventional balance training in subjects with subacute stroke.

Study 2: The purpose of this study was to investigate the effects of telerehabilitation with group therapy on balance and daily activities in subjects with stroke living in long-term care facilities (LTC).The null hypothesis would be telerehabilitation balance training were not significantly different from conventional balance training in subjects with subacute stroke.

study 3:To investigate whether a four-week tele-rehabilitation program can result in significant improvements in physical function and quality of life for subjects with chronic stroke living in long-term care facilities.

Study 4: To compare the effects of a home-based telerehabilitation (Tele) with intelligent agent systems and a conventional in-home physical therapy (home PT) for subjects with stroke.

DETAILED DESCRIPTION:
Study 1: Methods-Twenty-four subjects with substroke (less than 6 months post-stroke) were recruited for telerehabilitation group and conventional balance training group. Study 2. Methods-Twenty -four participants with mild to moderate stroke were randomized into telerehabilitation (Tele) group and conventional (Conv) group. They received balance training with three sessions per week for 4 weeks. The pressure distribution of buttock-pressure interface was measured by Pressure Distribution Plate (PDM-S).

Study 3.Methods: Twenty-four participants were recruited from three long-term care facilities. Participants were assigned into tele-rehabilitation (Tele group) and conventional Groups (Con group) randomly. Baseline and post-treatment physical function, daily activities and health-related quality of life (HRQOL) were assessed by Simplified-STREAM, Berge Balance scale (BBS), Barthel index (BI), and Stroke Impact Scale (SIS 3.0), respectively. Interventions were conducted to both groups by two different physical therapists with three sessions a week for four weeks of intervention.

Study 4. Ten participants with stroke were randomized into Tele or control group 1 (CG1) for randomized controlled trial. The Tele group also received home PT at 3 weeks later as control group 2 (CG2) for cross over design.

Intervention: All three groups received 4 weeks training (2 sessions/week, 50 minutes/session), including upper extremity and balance exercises.

Main outcome measures: The assessments were performed at baseline (pre), after 4 weeks (post) and after 7 weeks (follow-up). The measures for physical function included Stroke Rehabilitation Assessment (STREAM), Postural Assessment Scale for Stroke Patients (PASS), and Barthel index (BI). The measures for satisfaction included Stroke Impact Scale (SIS) and user-satisfaction questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Having a first episode of unilateral stroke with hemiparesis,
* Brunnstrom score between stages II and VI for the upper and lower hemiplegic extremities,
* Being able to understand and follow simple verbal instructions.

Exclusion Criteria:

* Those with other major diseases (e.g., Parkinson disease and severe osteoarthritis) and unstable medical conditions during the study period.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Changes of Berg Balance Scale | 1 month
  To measure static and dynamic balance during daily activities

SECONDARY OUTCOMES:
Changes of Stroke Impact Scale (SIS) | 1 month
  the quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Hwa Lin, PhD, Principal Investigator — School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan